CLINICAL TRIAL: NCT04814511
Title: Prospective, Open-label, Multicenter, Initially Single-armed and in Case of Treatment Failure Subsequently Three-armed Randomized Clinical Trial of Phase III/IV Investigating the Escalated Therapy of Scabies With INFECTOSCAB 5% (Permethrin)
Brief Title: Escalated Therapy of Scabies With INFECTOSCAB 5% (Permethrin)
Acronym: ETSKABI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETSKABI; 2019-003234-16 (EudraCT Number)
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard therapy with InfectoScab 5 % Creme (Other)
  Interventions: Drug: InfectoScab 5 % Creme
- Escalated therapy with InfectoScab 5 % Creme (arm E5) (Experimental)
  Interventions: Drug: InfectoScab 5 % Creme
- Escalated therapy with Permethrin 10 % Creme (arm E10) (Experimental)
  Interventions: Drug: Permethrin 10 % Creme
- Escalated therapy with InfectoScab 5 % Creme in combination with Driponin 3 mg Tabletten (arm EK) (Experimental)
  Interventions: Drug: InfectoScab 5 % Creme; Drug: Driponin 3 mg Tabletten

INTERVENTIONS:
Drug: InfectoScab 5 % Creme — InfectoScab 5 % Creme is the already approved standard therapeutic agent, containing the active ingredient permethrin in 5 % concentration. In this study, it is used for topical treatment in the first treatment cycle (standard therapy) as well as in the second treatment cycle (escalation therapy).
  Arms: Escalated therapy with InfectoScab 5 % Creme (arm E5); Escalated therapy with InfectoScab 5 % Creme in combination with Driponin 3 mg Tabletten (arm EK); Standard therapy with InfectoScab 5 % Creme
Drug: Permethrin 10 % Creme — Permethrin 10 % Creme also contains permethrin as the active ingredient, but in 10 % concentration. Permethrin 10 % creme is used exclusively for topical treatment in the second therapy cycle (escalation therapy).
  Arms: Escalated therapy with Permethrin 10 % Creme (arm E10)
Drug: Driponin 3 mg Tabletten — Driponin 3 mg Tabletten are approved for the treatment of scabies, containing ivermectin as the active ingredient. Driponin is used as a supplementary, peroral add-on combination treatment in addition to topical permethrin therapy and is used exclusively in the second treatment cycle (escalation therapy).
  Arms: Escalated therapy with InfectoScab 5 % Creme in combination with Driponin 3 mg Tabletten (arm EK)

SUMMARY:
The ETSKABI study is a prospective, open-label, multicenter, initially single-armed and in case of treatment failure subsequently three-armed randomized clinical trial. Within the initial treatment phase, the to-date clinical efficacy of the standard therapy regimen according to the current German "S1-guideline for the diagnosis and treatment of scabies" is to be examined. The subsequent second phase focusses on three differently escalated treatment regimens in order to evaluate their potential to cure those patients still suffering from Scabies after standard therapy.

In total, 183 patients with Scabies who meet all inclusion criteria and do not meet none of the exclusion criteria are to be enrolled and topically treated with Permethrin 5 % cream (up to two administrations, i.e. repeated one-time on day 14 in case of persisting Scabies). In case of treatment failure by the end of phase one, adult patients will be randomized to either receive an (i) escalated therapy with Permethrin 5 % cream (repeated topical administration on two consecutive days), (ii) an add-on-combination consisting of escalated therapy with Permethrin 5 % cream and Ivermectin p.o. or (iii) an escalated therapy with Permethrin 10 % cream (up to two administrations, i.e. repeated one-time on day 14 in case of persisting Scabies).

The primary objective of the ETSKABI study is the clinical efficacy of the standard therapy by the end of phase one (standard therapy according to the S1-guideline). Beside this, clinical efficacy by the end of phase two (escalation phase) will be evaluated as well as adverse events in order to investigate over-all clinical safety.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute scabies disease: detection of mites and/or mite nymphs and/or mite larvae at scabies-typical predilection sites, detected by reflected light microscopy (dermatoscopy) or light microscopy of skin samples.
* Age between 6 and 85 years
* Written informed consent of the study participant (if of age) or of all guardians (in the case of study participants who are minors < 12 years of age) or of all guardians and the study participant (in the case of study participants who are minors ≥ 12 years of age).

Exclusion Criteria:

* Previous treatment with antiscabiosa in the last 14 days.
* Known intolerance to permethrin, other pyrethroids, chrysanthemum, ivermectin or any of the other ingredients of the study medication.
* Scabies crustosa
* Impetiginisation/eczematisation requiring in-patient treatment
* Body weight > 120 kg
* Pregnancy, lactation
* Immunodeficiency (of any kind, including extensive local therapy (>20% body surface area) with corticosteroids >2 weeks in the last 4 weeks or ≥ 10 mg prednisolone equivalent >7 days in the last 4 weeks- even without signs of scabies crustosa)
* Other serious illnesses which, in the opinion of the investigator, prevent the patient from participating in the study (including risk factors for severe COVID-19 disease in the case of SARS-CoV-2 infection).
* Planned systemic use of corticosteroids
* Planned or previous (last 4 weeks) use of systemic or cutaneous non-steroidal immunosuppressants
* Known or clinically suspected blood-brain barrier disruption (e.g. ABCB-1 (=MDR-1) mutation), and history of neurotoxic effects from ivermectin or other substrates/inhibitors of para-glycoprotein (P-gp)
* Apparent unreliability or unwillingness to cooperate.
* Inability to understand and comply with study instructions
* Known alcohol, medication or drug dependence
* Court/agency-ordered institutionalisation
* Dependence on sponsor or investigator
* Previous participation in a clinical trial within the last 30 days or in the same clinical trial

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Yes/No) | day 0 - day 28
  Efficacy (Yes/No) after completed standard therapy treatment cycle (InfectoScab 5 % Creme, up to two administrations, if necessary), i.e. treatment success on day 14 (one administration) or on day 28 (one readministration due to persisting Scabies on day 14).
  Treatment success is defined as:
  * absence of new scabietic skin lesions, AND
  * all remaining scabietic lesions are in healing, AND
  * exclusion of mite infestation in all non-healed efflorescences by reflected light microscopy (dermatoscope), possibly confirmed by microscopic examination of a skin sample, AND
  * exclusion of the usage of other anti-scabietic drugs

SECONDARY OUTCOMES:
Efficacy (treatment success) for VS1 and VS2, as well as for the corresponding follow-up visits FUS1 and FUS2 (separately and cumulatively). | day 14 - day 70
Efficacy (therapy success) for VE5, VE101/2 (separately and cumulatively) and VEK as well as for the corresponding follow-up visits FUE5/E10/EK, separately as well as cumulatively according to visit type (regular visit, FU visit) | day 28 - day 70
Cumulative efficacy (treatment success) of permethrin-only treatment (i.e. without combined escalation permethrin + ivermectin) by visit type (regular visit, FU visit) | day 28 - day 56
Frequency of required repeated standard therapy as well as escalated therapy. | day 0 - day 70
Itch (numerical rating scale (NRS) of 0-10) and change in itch vs baseline (scale differences) for all visits, for standard therapy and escalated therapy, and for escalated therapy additionally the change in itch vs start of escalated therapy. | day 0 - day 70
Number and type of body regions affected (wrists/hands, arm pouches, armpits, genital region, groin, knee, feet/ankles/lower legs, head, torso, other) for all visits. | day 0 - day 70
Proportion of patients (in %) with evidence of mites (incl. nymphs and larvae, reflecting light microscopy (dermatoscope) or light microscopy of skin samples) for all visits, for standard therapy and escalated therapy | day 0 - day 70
Proportion of patients with use of antiscabiosa not conforming to study procedures for all visits, for standard therapy and escalated therapy | day 0 - day 70
Proportion of patients with new scabies efflorescences for all treatment cycles and control visits | day 0 - day 70
Patients with "additionally confirmed" therapy failure (in %) | day 0 - day 70
  Proportion of patients with new scabies efflorescences at the end of standard therapy or escalated therapy OR with mite detection by microscopic examination of a skin sample at the aforementioned time points OR use of other antiscabiosa not conforming to the study procedure during the respective therapy cycle.
Patients with reinfestation (in %): Proportion of patients with microscopically confirmed new efflorescences at the end of standard therapy or escalated therapy (respective FU-visit) who were assessed as cured at the immediately preceding control visit. | day 0 - day 70
Adverse events, serious adverse events, unexpected drug reactions, serious unexpected drug reactions (total frequency, type, severity, causality, with frequencies, with separate presentation of local reactions). | day 0 - day 70

CONTACTS AND LOCATIONS:
Overall Officials: Cord Sunderkötter, Prof. Dr., Principal Investigator — Universitätsklinik und Poliklinik für Dermatologie und Venerologie
Locations (8):
- Germany (8):
  - Uniklinik RWTH Aachen, Aachen
  - Universitätsklinikum Augsburg, Augsburg
  - Klinikum Darmstadt, Darmstadt
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinik und Poliklinik für Dermatologie und Venerologie, Halle
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No